CLINICAL TRIAL: NCT07246083
Title: Study on Let's Talk
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Evidence and Implementation Singapore Ltd (Other)
Collaborators: MOH Office for Healthcare Transformation (MOHT), Singapore (Unknown)
Responsible Party: Principal Investigator, Jean Liu, Associate Director, Centre for Evidence and Implementation Singapore Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NUS-IRB-2025-151
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Mental Health Help-Seeking
Keywords: digital mental health

STUDY DESIGN:
Intervention Model Description: This intervention has several components:
  Experience sampling: During the 21-day experience sampling period, prompts will be sent at regular intervals during the waking hours of the day (approx 3-4 times in a day).These prompts will be delivered through participants' own mobile devices (e.g. through a WhatsApp, Facebook, or Telegram chatbot).
  Monitoring: At each prompt, participants will be asked to complete the 6-item state scale of the short-form Spielberger State-Trait Anxiety Inventory (STAI) asking participants how calm, tense, upset, relaxed, content, and worried they feel (rating of 1='not at all' and 4='very much').
  If participants report feeling 'moderately' or 'very much' anxious, they will then receive one of the following prompts (at random): (a) instructions to carry out an activity on the Let's Talk site (e.g., post a question to a therapist, post a question to peers, read prior responses), or (b) no further prompt. 30 minutes later, they will then be asked again: (
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ESM (Experimental): During the 21-day experience sampling period, prompts will be sent at regular intervals during the waking hours of the day (approx 3-4 times in a day).These prompts will be delivered through participants' own mobile devices (e.g. through a WhatsApp, Facebook, or Telegram chatbot). At each prompt, participants will be asked to complete the 6-item state scale of the short-form Spielberger State-Trait Anxiety Inventory (STAI) asking participants how calm, tense, upset, relaxed, content, and worried they feel (rating of 1='not at all' and 4='very much').
  If participants report feeling 'moderately' or 'very much' anxious, they will then receive one of the following prompts (at random): (a) instructions to carry out an activity on the Let's Talk site (e.g., post a question to a therapist, post a question to peers, read prior responses), or (b) no further prompt. 30 minutes later, they will then be asked again: (i) for their STAI ratings, and (ii) whether they had used the Let's Talk site.
  Interventions: Behavioral: let's talk forum

INTERVENTIONS:
Behavioral: let's talk forum — The platform also features an "Ask-a-Therapist" function, allowing users to anonymously pose questions to a panel of verified psychotherapists and receive a response within 24 hours. As such, Let's Talk provides a valuable case study to:
  * assess the real-time impact of digital peer support and professional input, and
  * explore how anonymous online interactions may support emotion regulation and enhance well-being

SUMMARY:
The goal of this experience sampling method study is to understand the effectiveness and user experience of the 'let's talk' forum-- a public platform designed by the Ministry of Health Office for Healthcare Transformation (MOHT) to provide just-in-time digital mental health support for youths. 'Let's Talk' is a joint initiative by MOHT, Ministry of Social and Family Development (MSF), National Council of Social Service (NCSS), and the Institute of Mental Health (IMH) in Singapore.

Participants who meet the eligibility criteria (based on DASS-21 cutoff scores) will be invited to participate in Phase 2, which involves a 21-day intervention period involving the 'let's talk' forum. The experience sampling protocol involves sending prompts at regular intervals and monitoring anxiety levels.

DETAILED DESCRIPTION:
This study will involve three phases: (a) screening / baseline, (b) experience sampling, and (c) focus group discussions. Recruitment: Participants will be recruited through a combination of targeted and public outreach strategies. For non-NUS students, recruitment posters will be disseminated online via platforms such as Research Lobang, partner mailing lists, the study team's personal and professional social media accounts, and through a snowball sampling approach. Partner mailing lists will include those from our collaborating organisations, limited to participants who have consented to receive email communications. For National University of Singapore (NUS) students, pending relevant institutional approvals, recruitment posters will be shared through departmental email lists and social media platforms, targeting departments such as Psychology, Medicine, Science, and Engineering. Interested individuals will be directed to an online sign-up link included in the advertisement. Upon expressing interest, they will receive a link to a screening survey hosted on Qualtrics. Email invitations will be sent by authorised personnel with permissions to use the mailing list. We will also share the advertisement materials with MOHT who may assist in amplifying outreach to participants engaged through their previous campaigns or partner initiatives (excluding MOHT employees). Only participants who have consented to be contacted will be reached out to.

Phase 1: Screening Participants will sign up by responding to an online link provided in the advertisements. They will then be provided a survey link hosted on Qualtrics.

After reading a participant information sheet and providing consent, participants will complete questions on:

* Mental health symptoms: Measured through the 21-item Depression, Anxiety and Stress Scale (DASS-21);
* Awareness, views and prior usage of mental health services, including let's talk, digital mental health services, and other mental health services. As part of this series of questions, they will be asked to complete the 10-item Attitudes Toward Seeking Professional Psychological Help Scale - Short Form (ATSPPH-SF); and
* Demographics.

Phase 2: Experience sampling method protocol Participants who meet the eligibility criteria (based on DASS-21cutoff scores, see inclusion criteria section) will be invited to participate in Phase 2, which involves a 21-day intervention period on the let's talk forum.

1. Briefing and baseline measures At the start of the study, participants will be introduced to the let's talk platform and the study overview through a briefing handout and/or an online briefing session.

   They will also be asked to complete the following measures:
   * Attitudes, knowledge and behaviors regarding mental health and help-seeking: 28-item Stigma Scale, the 35-item Mental Health Literacy Scale (MHLS), and the 9-item Mental Help Seeking Attitudes Scales (MHSAS).
   * Emotion regulation: 28-item Coping Orientation to Problems Experienced Inventory (Brief-COPE) and 18-item Difficulties in Emotion Regulation Scale (DERS-18)
   * Sense of isolation/belonging: 10-item UBC State Social Connection Scale (UBC-SSCS)
2. let's talk intervention Unlike appointment-based counselling services, online mental health forums offer users the promise of 'just-in-time' service delivery that: (a) is available 24/7, and (b) can address mental health needs as and when they arise.

   Despite the 'just-in-time' nature of these platforms, little is known about the real-time impact of forum-based services. Accordingly, we plan to run an experience sampling study to introduce and monitor the intervention.

   This intervention has several components:
   * Experience sampling: During the 21-day experience sampling period, prompts will be sent at regular intervals during the waking hours of the day (approx 3-4 times in a day).These prompts will be delivered through participants' own mobile devices (e.g. through a WhatsApp, Facebook, or Telegram chatbot).
   * Monitoring: At each prompt, participants will be asked to complete the 6-item state scale of the short-form Spielberger State-Trait Anxiety Inventory (STAI) asking participants how calm, tense, upset, relaxed, content, and worried they feel (rating of 1='not at all' and 4='very much').

   If participants report feeling 'moderately' or 'very much' anxious, they will then receive one of the following prompts (at random): (a) instructions to carry out an activity on the Let's Talk site (e.g., post a question to a therapist, post a question to peers, read prior responses), or (b) no further prompt. 30 minutes later, they will then be asked again: (i) for their STAI ratings, and (ii) whether they had used the Let's Talk site.

   - If participants report feeling low anxiety ('not at all' or 'somewhat'), they will receive no further prompt.

   As per typical ESM protocols, they will have a 30-minute window to respond. If they fail to respond during that window, it will be logged as a non-response.

   Should participants choose to respond to our prompts and use the let's talk site, this will occur anonymously and will be independent from the study. (We will not be tracking participants' use of the let's talk site directly.)

   Globally, the typical experience sampling protocol is 7 times a day for all days. In our previous experiments, participants had no objections to being contacted 3-4 times a day. At any point of time, participants can choose to drop out from the study at will.
3. Follow up measures

Immediately after the intervention and one month later, participants will be asked a combination of the following measures:

* Mental health symptoms: Measured through the 21-item Depression, Anxiety and Stress Scale (DASS-21);
* Awareness, views and use of mental health services during the interim period, including digital mental health services and other mental health services. As part of this series of questions, they will be asked to complete the 10-item Attitudes Toward Seeking Professional Psychological Help Scale - Short Form (ATSPPH-SF); and
* Attitudes, knowledge and behaviors regarding mental health and help-seeking: 28-item Stigma Scale, the 35-item Mental Health Literacy Scale (MHLS), and the 9-item Mental Help Seeking Attitudes Scales (MHSAS).
* Emotion regulation: 28-item Coping Orientation to Problems Experienced Inventory (Brief-COPE) and 18-item Difficulties in Emotion Regulation Scale (DERS-18)
* Sense of isolation / belonging: 10-item UBC State Social Connection Scale (UBC-SSCS)
* Feedback on the Let's Talk site: Participants will be asked to provide feedback the site (e.g., continued usage of site, usage outside the prompts, perceived utility of each feature).

Majority of the forum, including the responses is publicly accessible. Participants are treated like regular users on the platform and employees will know not that they are a research participant.

Participants who self-report very high levels of distress are not ignored at any stage. If they report high distress, they will receive prompts directing them to evidence-based resources available on the platform, including clear information on how and where to seek professional help if needed. At the 30-minute follow-up, if participants continue to indicate very high distress (or if they do not respond), they will again be directed to these resources and reminded of available professional support options, including speaking with a therapist on the site. This ensures that participants consistently receive guidance and are encouraged towards appropriate help-seeking rather than left unsupported.

Phase 3: Focus group discussions (FGDs)

In Phase 3, we will conduct focus group discussions with:

* Participants from Phase 2 who have completed the Phase 2 components and are interested in joining focus group discussions, and
* Existing befrienders / peer support leaders on the Let's Talk site. For phase 3 recruitment, MOHT will reach out to their network of peer supporters and befrienders.

The FGDs will be conducted online (Eg: Zoom or Microsoft Teams) They will be audio and video recorded and transcribed for research purposes. With participant consent, quotes from the FGDs may be used anonymously in publications and presentations. Although only the audio recording is required for transcription, the online application's automatic recording feature will be used for convenience, resulting in a video recording as well. The video will be used solely to verify observations or match speaker names in the transcript before being deleted.

A team of trained facilitators will be scheduled to lead the sessions, depending on availability and group composition.

To maintain participants' privacy, all participants will be encouraged to turn off their cameras during the FGDs. Researchers will also provide instructions on how to change their display name on Zoom/Teams to something anonymous, and will remind participants of this option at the start of each session. These steps aim to ensure a safe and confidential space for open sharing.

10 participants from phase 2 and 10 befrienders from the platform. 2-4 FGDs in total 1 hour each. (1 or 2 FGD per group)

FGDs will focus on implementation, effectiveness and peer supporter themes. The questions asked during the FGDs cover the following themes (see interview guide attached, detailed guide will be attached through a future modification)

* What are the barriers and enablers to accessing and returning to Let's Talk?
* To what extent have the key features of let's talk been accessed?
* To what extent have let's talk showed evidence that the intended goals were realised?
* What was the impact on users?
* What was the impact on peer supporters?

ELIGIBILITY:
Phase 1 Screening Inclusion Criteria:

* Aged between 18-25 years if they are a student at the National University of Singapore (NUS); 21-25 years old if they are not a student at NUS
* Must have lived in SG for at least 2 years
* Have not received a formal diagnosis of a psychiatric disorder
* Not currently receiving any form of mental health treatment (e.g., counselling)

Phase 2 Experience Sampling Inclusion Criteria:

- Partiicpants from Phase 1 whose DASS-21 scores are at least moderate for any one of the following sub scales (cut off of 14 for depression, 10 for anxiety, and 19 for stress).

Phase 3 Focus Group Discussions Inclusion Criteria:

* Existing befrienders or peer supporters on the let's talk site (aged 21-80)
* Agree to audio and video recording of FGD
* Individuals who have completed phase 2

Exclusion Criteria:

* Those who do not meet the inclusion criteria will be screened and excluded.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Mental health symptoms: Measured through the 21-item Depression, Anxiety and Stress Scale (DASS-21) | Screening
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest / involvement, anhedonia and inertia. The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The stress scale is sensitive to levels of chronic non-specific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset / agitated, irritable / over-reactive and impatient. Scores for depression, anxiety and stress
Awareness, views and prior usage of mental health services | Screening, 4 weeks after baseline, 8 weeks after baseline
  As part of this series of questions, they will be asked to complete the 10-item Attitudes Toward Seeking Professional Psychological Help Scale - Short Form (ATSPPH-SF). The ATSPPH-SF is a 10-item measure used to assess ATSPPH on a 4-point Likert scale, ranging from 0 to 3. Higher total score indicates more positive ATSPPH and is associated with lower levels of stigma against mental illness (Elahi et al., 2008). The ATSPPH-SF was reported to have unidimensional structure with Cronbach's alpha values of 0.84. Construct validity was reported to be 0.87, which was estimated by correlating it with the longer version (Fischer & Farina, 1995).
Attitudes, knowledge and behaviors regarding mental health and help-seeking | Baseline, 4 weeks after baseline, 8 weeks after baseline
  The Mental Health Literacy Scale (MHLS) is a 35-item, scale-based measure of knowledge and beliefs about mental disorders which aid their recognition, management or prevention (Jorm et al., 1997; O'Connor & Casey, 2015). The MHLS assesses six attributes of mental health literacy.
STAI Rating | Daily over 21 days
  The Spielberger State-Trait Anxiety Inventory (STAI) 6-item form is a shortened version of the original STAI, developed by Marteau and Bekker in 1992, which uses six items to measure state anxiety (how a person feels at the moment) while reducing respondent burden. This shorter scale maintains acceptable reliability and validity, produces scores comparable to the full-form, and is sensitive to fluctuations in anxiety.
Emotion Regulation | 4 weeks after baseline, 8 weeks after baseline
  The Brief-COPE is a 28 item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event.
Attitudes, knowledge and behaviors regarding mental health and help-seeking | Baseline, 4 weeks after baseline, 8 weeks after baseline
  MHSAS is a survey about mental health seeking attitudes, using a seven-point scale. It has nine items and produces a single mean score.
Emotion regulation | 4 weeks after baseline, 8 weeks after baseline
  DERS-18 is a brief version of the Difficulties in Emotion Regulation Scale, with 18 items, and is a brief version of the original 36 item DERS.

SECONDARY OUTCOMES:
Sense of isolation/belonging using UBC-SSCS | Baseline, 4 weeks after baseline, 8 weeks after baseline
  The UBC State Social Connection Scale (UBC-SSCS) is a 10-item scale developed to measure momentary feelings of social connection.
Feedback on the let's talk forum | 4 weeks after baseline, 8 weeks after baseline
  Participants will be asked to provide feedback on the site such as continued usage of site, usage outside the prompts, perceived utility of each feature.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Liu, Principal Investigator — Centre for Evidence and Implementation
Locations (2):
- Singapore (2):
  - National University of Singapore, Singapore, Singapore
  - National University of Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saw YE, Tan EY, Liu JS, Liu JC. Predicting Public Uptake of Digital Contact Tracing During the COVID-19 Pandemic: Results From a Nationwide Survey in Singapore. J Med Internet Res. 2021 Feb 3;23(2):e24730. doi: 10.2196/24730. PMID 33465034
- [Background] Tan EY, Wee RR, Saw YE, Heng KJ, Chin JW, Tong EM, Liu JC. Tracking Private WhatsApp Discourse About COVID-19 in Singapore: Longitudinal Infodemiology Study. J Med Internet Res. 2021 Dec 23;23(12):e34218. doi: 10.2196/34218. PMID 34881720
- [Background] Barsova T, Cheong ZG, Mak AR, Liu JC. Predicting Psychological Symptoms When Facebook's Digital Well-being Features Are Used: Cross-sectional Survey Study. JMIR Form Res. 2022 Aug 29;6(8):e39387. doi: 10.2196/39387. PMID 36036971
- [Background] Erdembileg, S., Asplund, C. L., & Liu, J. C. J. (in preparation). Engagement with Taylor Swift's music and social media content predicts mental health outcomes in youths: Cross-sectional survey study.